CLINICAL TRIAL: NCT02630875
Title: An Exploratory Phase II Study to Demonstrate the Safety and Efficacy of A4250 in Children With Cholestatic Pruritus
Brief Title: A4250, an IBAT Inhibitor in Pediatric Cholestasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albireo (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4250-003
Record Dates: First submitted 2015-11-23; First posted 2015-12-15 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Pediatric Cholestasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- A4250 1 (Active Comparator): Dose I
  Interventions: Drug: A4250
- A4250 2 (Active Comparator): Dose 2
  Interventions: Drug: A4250
- A4250 3 (Active Comparator): Dose 3
  Interventions: Drug: A4250
- A4250 4 (Active Comparator): Dose 4
  Interventions: Drug: A4250
- A4250 5 (Active Comparator): Dose 5
  Interventions: Drug: A4250
- A4250 6 (Active Comparator): Dose 6
  Interventions: Drug: A4250

INTERVENTIONS:
Drug: A4250 — A4250

SUMMARY:
This study will evaluate A4250 (IBATinhibitor) as a treatment option in pediatric patients with chronic cholestasis with main emphasis on safety evaluation and on effects on pruritus

DETAILED DESCRIPTION:
The primary aims of this Phase II exploratory study in patients treated with A4250 due to cholestasis induced pruritus are to:

* Assess the safety and tolerability of A4250, orally administered first as a single dose and then during a four week treatment period, as determined by the occurrence of treatment-emergent SAEs
* Explore changes in serum total bile acids after a four week treatment period

Secondary safety aims include assessment of the safety and tolerability of A4250, orally administered first as a single dose and then during a four week treatment period, as determined by the occurrence of treatment-emergent AEs and changes in safety parameters including laboratory tests and vital signs

Secondary efficacy aims are to:

* Demonstrate the efficacy of A4250, orally administered during a four week treatment period, on liver biochemistry variables and on pruritus parameters
* Evaluate the pharmacokinetic properties of A4250 orally administered first as a single dose and then after a four week treatment period
* Evaluate changes in VAS-itching score after a four week treatment period

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pruritus due to chronic cholestasis based on history and investigator judgment. This will include but will not be restricted to patients with Progressive familial intrahepatic cholestasis (PFIC), Alagille syndrome (ALGS), Biliary Atresia and Sclerosing Cholangitis

Exclusion Criteria:

* Any condition that in the opinion of the investigator constitutes a risk for the patient or a contraindication for participation and completion of the study, or could interfere with study objectives, conduct, or evaluations
* Clinical or biochemical signs of decompensated liver disease
* Liver transplantation

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08; Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
AE evaluation | 4 wks
  Treatment-emergent SAEs Adverse events

SECONDARY OUTCOMES:
Bile acid changes | 4 weeks
  Evaluation of bile acids

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (7):
- Department of Pediatric and Adolescent Medicine Rigshospitalet, Copenhagen, Denmark
- France (2):
  - Pediatric Hepatology and Liver Transplantation, University Hospitals of Paris-Sud, Paris, Orsay
  - Department of Pediatric Gastroenterology Hepatology-Nutrition, Necker-Enfants maladies hospital, Paris
- Germany (2):
  - Pediatric Gastroenterology and Hepatology, Pediatric Surgery, Hannover, Hanover
  - Gastroenterology/Hepatology, University Hospital for Children and Adolescents, Tübingen
- Henrik Arnell, Stockholm, Sweden
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants. Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/